CLINICAL TRIAL: NCT00234390
Title: Prevention of Asthma in Infants/Young Children - PAC
Brief Title: PreAsthmaControl (PAC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-004-0299
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

INTERVENTIONS:
Drug: Pulmicort (budesonide) pMDI

SUMMARY:
The purpose of this study is to investigate the ability of budesonide, given during episodes of troublesome lung symptoms to reduce further symptoms in infants and young children at risk of developing asthma

ELIGIBILITY:
Inclusion Criteria:

* Children of asthmatic mothers form the COPSAC birth cohort study

Exclusion Criteria:

* Children born more than 4 weeks preterm
* children with other systemic illness that atopy/allergy
* Children requiring mechanical ventilation at any time since birth.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Start 1998-11; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
symptom free days
days with no use of bronchodilator
days with no use of bronchodilator and no symptoms
number of treated episodes
number of treatment with add-on medication

SECONDARY OUTCOMES:
asthma status
time to start of algorithm treatment
the total steroid dose
First treatment episode:
number of symptom days
number of days with use of bronchodilator
number of patients who needed add-on medication
BMD
height
serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AB CNS Medical Science Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Copenhagen, Denmark

REFERENCES:
- [Result] Bisgaard H, Hermansen MN, Loland L, Halkjaer LB, Buchvald F. Intermittent inhaled corticosteroids in infants with episodic wheezing. N Engl J Med. 2006 May 11;354(19):1998-2005. doi: 10.1056/NEJMoa054692. PMID 16687712